CLINICAL TRIAL: NCT03498690
Title: Protocol Lab for Online Trials-Delphi (PLOT-D)
Brief Title: Protocol Lab for Online Trials-Delphi
Acronym: PLOT-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ThinkWell (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PLOT-D Ranking
Record Dates: First submitted 2018-04-01; First posted 2018-04-17 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Decisional Variability by Presentation Methods for Consensus
Keywords: online trial; decision analysis

STUDY DESIGN:
Intervention Model Description: Randomized 1:1:1 to feedback that is integrative or role specific or presented consecutively
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Integrative (Active Comparator)
  Interventions: Behavioral: Integrative
- Role Specific (Active Comparator)
  Interventions: Behavioral: Role specific
- Consecutive (Active Comparator)
  Interventions: Behavioral: Consecutive

INTERVENTIONS:
Behavioral: Integrative — Stakeholder groups: a-b
  Arms: Integrative
Behavioral: Role specific — Stakeholder groups: a or b
  Arms: Role Specific
Behavioral: Consecutive — Stakeholder groups: a=> b
  Arms: Consecutive

SUMMARY:
The Protocol Lab for Online Trials-Delphi (PLOT-D) module will use an online three-round Delphi combined with Participatory action research to inform the development of a multi-use protocol template to use in writing protocols for self-recruited online trials of interventional self-management. The Delphi will include an embedded randomized controlled trial to test how and if stakeholders adapt their views based on the contributions of others inside or outside the groups with which they are familiar.

DETAILED DESCRIPTION:
The research aims to provide support for citizens to work alongside researchers to build participatory health trials online (any randomized trial that uses the internet for a health or wellness intervention). Tools to develop methods to run quality online trials protocols are needed. Also, help for adapting guidance to include the public and patients as partners in research for online trials is limited. The purpose of this work is to facilitate improved practice within protocol writing for participatory online trials.

Public and patient involvement (PPI), is one method used to conduct participatory research. PPI actively engages communities or individuals and moves beyond educating, engaging or doing interviews with research participants and does the research with them as partners. There is growing consensus that PPI is of value to researchers, industry, regulators, and members of the public.

There is an active discussion that is without substantial evidence for when the optimal time in the research process is to start PPI and whether patients and the public should join the research team, act as advisors, or have everyone contribute perspectives and work with their roles or peer groups.

The embedded study within the Delphi explores how working with stakeholder feedback in different ways may influence decision ranking as well choice similarities and differences

ELIGIBILITY:
Inclusion Criteria:

* Protocol lab for online trials Delphi (PLOT-D) participants

Exclusion Criteria:

* None if inclusion criteria are met

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
The top five disparities and similarities in ranking between interventions | Up to 20 weeks or study completion
  Prioritization of method preferences as decided by participants

SECONDARY OUTCOMES:
Differences and similarities between stakeholder groups | Up to 20 weeks or study completion
  Ranking differences between stakeholders randomized to different forms of information presentation

CONTACTS AND LOCATIONS:
Overall Officials: Amy I Price, PhD, Principal Investigator — University of Oxford; Mike J Clarke, DPhil, Principal Investigator — Queen's University, Belfast
Locations (1):
- ThinkWell, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Aggregated de-identified data will be available on request to principal investigator Amy Price dr.amyprice@gmail.com
Supporting Information: Study Protocol, ICF
Time Frame: following publication and for 5 years
Access Criteria: email investigator dr.amyprice@gmail.com

REFERENCES:
- [Background] Sinha IP, Smyth RL, Williamson PR. Using the Delphi technique to determine which outcomes to measure in clinical trials: recommendations for the future based on a systematic review of existing studies. PLoS Med. 2011 Jan 25;8(1):e1000393. doi: 10.1371/journal.pmed.1000393. PMID 21283604
- [Background] Fletcher AJ, Marchildon GP. Using the Delphi Method for Qualitative, Participatory Action Research in Health Leadership. International Journal of Qualitative Methods 2014;13:1-18
- [Background] Brice A, Price A, Burls A. Creating a database of internet-based clinical trials to support a public-led research programme: A descriptive analysis. Digit Health. 2015 Nov 20;1:2055207615617854. doi: 10.1177/2055207615617854. eCollection 2015 Jan-Dec. PMID 29942546
- [Background] Bagley HJ, Short H, Harman NL, Hickey HR, Gamble CL, Woolfall K, Young B, Williamson PR. A patient and public involvement (PPI) toolkit for meaningful and flexible involvement in clinical trials - a work in progress. Res Involv Engagem. 2016 Apr 27;2:15. doi: 10.1186/s40900-016-0029-8. eCollection 2016. PMID 29062516
- [Background] Snow R, Crocker JC, Crowe S. Missed opportunities for impact in patient and carer involvement: a mixed methods case study of research priority setting. Res Involv Engagem. 2015 Aug 4;1:7. doi: 10.1186/s40900-015-0007-6. eCollection 2015. PMID 29062496
- [Background] Price A, Albarqouni L, Kirkpatrick J, Clarke M, Liew SM, Roberts N, Burls A. Patient and public involvement in the design of clinical trials: An overview of systematic reviews. J Eval Clin Pract. 2018 Feb;24(1):240-253. doi: 10.1111/jep.12805. Epub 2017 Oct 27. PMID 29076631